CLINICAL TRIAL: NCT01547897
Title: A Phase IIa Study to Characterize the Effects of CCL2 Inhibition With the Spiegelmer® NOX-E36 in Patients With Type 2 Diabetes Mellitus and Albuminuria
Brief Title: NOX-E36 in Patients With Type 2 Diabetes Mellitus and Albuminuria
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: TME Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SNOXE36C301; 2011-005710-11 (EudraCT Number)
Record Dates: First submitted 2012-02-27; First posted 2012-03-08 (Estimated); Last update posted 2014-02-24 (Estimated); Status verified 2013-09

CONDITIONS: Type 2 Diabetes Mellitus; Albuminuria
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Albuminuria

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- NOX-E36 (Active Comparator)
  Interventions: Drug: NOX-E36
- Placebo (Placebo Comparator)
  Interventions: Drug: NOX-E36

INTERVENTIONS:
Drug: NOX-E36 — 0.5 mg/kg study drug or placebo as SC injections twice a week

SUMMARY:
Primary objective:

- To characterize the effects of 12 weeks treatment with study drug on albumin-creatinine ratio (ACR) in patients with type 2 diabetes and albuminuria

Secondary objectives:

* To characterize the effect of study drug on glycosylated hemoglobin fraction (HbA1c)
* To evaluate the effect of study drug on markers of glycemic disorders, systemic inflammation, renal and liver disease and cardiovascular function
* To assess the safety and tolerability of study drug
* To determine the population pharmacokinetics (PK) of study drug

ELIGIBILITY:
Inclusion Criteria:

1. Type 2 diabetes mellitus according to American Diabetes Association (ADA) definition
2. Age ≥ 18
3. HbA1c between 6.0% and 10.5%, inclusive
4. ACR > 100 mg/g calculated 3 times in first morning void urine, at least 2 of the measurements > 100 mg/g
5. Patients on stable (unchanged medication for at least 3 months) treatment to control hypertension, hyperglycemia and (if applicable) dyslipidemia
6. Stable treatment with angiotensin-converting enzyme inhibitors (ACEi) and/or Angiotensin II receptor blockers (ARBs) (renin-angiotensin system [RAS] blockade)
7. Willing and able to understand and sign an approved Informed Consent form
8. Men must agree to follow accepted birth control methods during treatment and for 3 months after completion of treatment. Women must be of non-childbearing potential.

Exclusion Criteria:

1. Type 1 diabetes mellitus
2. Estimated Glomerular Filtration Rate (eGFR) ≤25 mL/min/1.73m2 (calculated by the Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI] formula)
3. Recent cardiovascular events (3 months)
4. Uncontrolled hypertension (upper limits 180/110 mmHg)
5. Dialysis and/or acute kidney injury within 3 months before screening
6. Significant edema, infectious diseases, leg ulcers
7. Severe concurrent disease which, in the judgment of the investigator, would interfere significantly with the assessments of safety and efficacy during this study
8. Treatment with any other investigational agent, or participation in another clinical study within 90 days prior to baseline visit
9. Patient with known infection with human immunodeficiency virus (HIV), Hepatitis B or Hepatitis C
10. In the judgment of the clinical investigator, clinically significant abnormal laboratory values at the screening visit
11. Use of thiazolidinedione class drugs, immune suppressants, steroid therapy (except for topical use or inhalation), chronic use of non-steroidal anti-inflammatory drug (NSAIDs), cyclooxygenase type 2 (COX-2) inhibitors, two or more diuretic drugs and/or aliskiren
12. In the judgment of the clinical investigator, patients who are likely to be non-compliant or uncooperative during the study.
13. Previous participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2012-03; Primary Completion 2013-09 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Effect of NOX-E36 on albuminuria as measured by ACR (albumin to creatinine ratio; mg/g) | Change versus baseline after 12 weeks treatment
  ACR calculated in first morning void urine; comparison of patients treated with NOX-E36 versus placebo

SECONDARY OUTCOMES:
Effect of NOX-E36 on hsCRP | Change versus baseline after 12 weeks treatment
  Comparison of patients treated with NOX-E36 versus placebo
Effect of NOX-E36 on HbA1C | Change versus baseline after 12 weeks treatment
  Comparison of patients treated with NOX-E36 versus placebo
Effect of NOX-E36 on HOMA-IR | Change versus baseline after 12 weeks treatment
  Comparison of patients treated with NOX-E36 versus placebo
Effect of NOX-E36 on eGFR | Change versus baseline after 12 weeks treatment
  eGFR will be calculated by the CKD-EPI equation using creatinine and cystatin C
  Comparison of patients treated with NOX-E36 versus placebo

CONTACTS AND LOCATIONS:
Overall Officials: Kai Riecke, MD, Study Director — Noxxon AG
Locations (24):
- Prague, Czechia
- Germany (10):
  - Aschaffenburg
  - Dortmund
  - Düsseldorf
  - Hanover
  - Kronberg
  - Mainz
  - Mannheim
  - Offenbach
  - Schwabenheim
  - Witten
- Hungary (6):
  - Balatonfüred
  - Budapest
  - Gyula
  - Miskolc
  - Pécs
  - Szeged
- Poland (4):
  - Bialystok
  - Grodzisk Mazowiecki
  - Katowice
  - Warsaw
- Romania (3):
  - Arad
  - Bucharest
  - Timișoara

REFERENCES:
- [Derived] Park EJ, Choi J, Lee KC, Na DH. Emerging PEGylated non-biologic drugs. Expert Opin Emerg Drugs. 2019 Jun;24(2):107-119. doi: 10.1080/14728214.2019.1604684. Epub 2019 Apr 19. PMID 30957581